CLINICAL TRIAL: NCT04206592
Title: A Prospective, Controlled and Randomized Comparison of the Ambu AuraGain and Intersurgical i-Gel Laryngeal Masks in Elective Laparoscopic Cholecystectomy
Brief Title: Comparison of the Ambu AuraGain and Intersurgical i-Gel Laryngeal Masks in Elective Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Plató (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MLA- Anesth
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2019-11

CONDITIONS: Airway Management; Laryngeal Masks
Keywords: Laryngeal mask; Oropharyngeal leak pressure; Laparoscopic Cholecystectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- i Gel LMA (Active Comparator): The sealing pressure of the igel laryngeal mask will be measured during pneumoperitoneum in elective laparoscopic cholecystectomy
  Interventions: Device: Oropharyngeal leak pressure during pneumoperitoneum.
- Ambu Aura Gain (Active Comparator): It will be compared the Ambu Aura Gain LMA vs iGel in elective laparoscopic cholecystectomy
  Interventions: Device: Oropharyngeal leak pressure during pneumoperitoneum.

INTERVENTIONS:
Device: Oropharyngeal leak pressure during pneumoperitoneum. — Oropharyngeal Leak Pressure (OLP) will be measured by closing the expiratory valve of the circle system at a fixed gas flow of 3 litres/min (maximum allowed 40 cmH2O) recording the pressure at which equilibrium has been reached or audible air is leaking.

SUMMARY:
Prospective, controlled, randomized study to compare Ambu AuraGain with Intersurgical i-Gel mask during mechanical ventilation in patients undergoing laparoscopic cholecystectomy.

The investigators hypothesise that when comparing the Ambu® AuraGainTM with Intersurgical i-GelTM mask, the Ambu® AuraGainTM would exhibit a higher oropharyngeal leak pressure (OLP) during mechanical ventilation in patients undergoing laparoscopic cholecystectomy.

The main goal is to compare the Ambu AuraGain with the i-Gel in terms of safety and efficacy during mechanical ventilation in critical phase of the pneumoperitoneum in lateral decubitus and reverse trendelemburg position. Secondary objectives are comparing insertion time, number of attempts, ventilatory airway peak pressure, time and success rates for gastric tube insertion and the incidence of side effects.

DETAILED DESCRIPTION:
Design: Prospective, controlled, randomized study. Participants: After approval by the local Clinical Research Ethics Committee, all patients scheduled for elective laparoscopic cholecystectomy at Hospital Plató (Barcelona) will be screened for participation. Patients will be informed about the study and they must provide written consent.

The need for orotracheal intubation during surgery will be considered as a study withdrawal criterion.

The primary outcome is the oropharyngeal leak pressure (OLP).

The secondary outcomes are: insertion time, number of attempts, ventilatory airway peak pressure, time, and success rates for gastric tube insertion and side effects.

Sample size has been calculated to detect a significant difference in oropharyngeal leak pressure (OLP) between two devices. According to the results of previous studies, the investigators assume a mean OLP of 29.2 (3.3) cmH2O for the i-Gel and of 34 (5) cmH2O for the Ambu AuraGain. In order to detect a difference of 10%, assuming a standard deviation of 5 cmH2O for both devices, 44 patients are required per group with a power of 80% and an alpha error of 0.05. To cover against a dropout rate of 10%, a total of 98 patients will be recruited.

The patients included in the study will be numbered consecutively and assigned to one of the two groups, 'LMA Ambu AuraGain' or 'i-gel', using a computer-generated random number table, by the principal investigator. The individual result will be kept in opaque envelopes. After the recruitment, the day of the procedure, the enrolling investigator will open sealed, opaque envelopes that conceal the group allocation. Participants will be blinded to their group allocation.

Procedures In the operating room, intravenous access will be secured and routine monitoring using ECG, non-invasive blood pressure, heart rate, oxygen saturation, end-tidal carbon dioxide (EtCO2) and sevoflurane (EtSevo) (Datex-Ohmeda S/5 Compact Critical Care Monitor; GE Healthcare). After pre-oxygenation with 100% oxygen by facemask for 3 min, anaesthesia will be induced with intravenous Fentanyl 50 μg/ml (2μg/kg), Propofol 1% (2-3 mg/kg) and Rocuronio 1% (0,6 mg/kg). The investigators will continue ventilating with 100% oxygen using a facemask at least for 1 min until optimum conditions for laryngeal mask insertion are achieved (loss of eyelash reflex, relaxation of the jaw, immobility, and apnoea).

Anesthesia will be maintained with Sevoflurane 2% in an air-oxygen mixture using a circle system with a fresh gas flow of 2 l/min. Additional intravenous Fentanyl will be administrated as clinically needed during anesthesia by an increase of 10-20% in blood pressure or heart rate. Laryngeal masks size will be determined according to the manufacturers weight-based recommendations and the insertion technique will be according to the recommendations of the Instruction Manual. After successful insertion, the cuff will be inflated with air until 60 cmH2O intracuff pressure (ICP) measured using an Ambu® airway pressure manometer (AMBU, S.L. B- 81040149, Alcala, Madrid, Spain). The second measurement of intracuff pressure will be performed for surgeries taking over an hour to ensure that the intracuff pressure has not changed significantly (± 5 cmH2O) since the last calibrated intracuff pressure. An effective airway will be judged by a square wave capnograph trace, bilateral chest auscultation and no audible leak with peak airway pressures at 12 cmH2O or greater during gentle manual ventilation. The device will be connected to the respiratory machine (Datex-Ohmeda S/5 Compact Critical Care Monitor; GE Healthcare) and patients will be ventilated with a tidal volume of 8 ml/kg, adjusting the respiratory rate to an end-tidal CO2 of 30-35mmHg.

A gastric tube will be inserted via the drain tube. The correct placement of the gastric tube will be confirmed by free movement during insertion and by aspiration of gastric fluid or detection of injected air by epigastric auscultation. Oropharyngeal Leak Pressure (OLP) will be measured by closing the expiratory valve of the circle system at a fixed gas flow of 3 liters/min (maximum allowed 40 cmH2O) recording the pressure at which equilibrium has been reached or audible air is leaking.

The leak pressure will be recorded before peritoneal insufflation and during pneumoperitoneum. The peritoneal insufflation pressure will be set at 12 mmHg. At the end of the surgery, the anesthesiologist will remove the laryngeal masks when the patients obey commands. The patients will be transferred to the Post-Anaesthesia Care Unit (PACU) to be monitored after the surgery.

Statistical Analysis Data will be entered into an Excel Database. All statistical analyses will be conducted using software from the Statistical Package for the Social Sciences (SPSS, Version 18.0, Chicago, IL, USA). The distribution of data will be determined using Kolmogorov- Smirnov analysis. The quantitative variables will be summarized with means and standard deviations or with medians and percentiles P25 and P75 in case of asymmetric distributions, and qualitative variables with frequencies and percentages. To study the relationships between qualitative variables, contingency tables will be made and the Chi-square or Fisher's tests will be used. The difference in oropharyngeal leak pressure (OLP) between two devices will be analyzed by a Student ́s t-test or the Mann-Whitney U test in case of non-normal distributions. To compare the incidence of side effects between the groups, the exact Fisher test or Chi-squared tests will be used. Significant differences will be quantified with 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 year
* American Society of Anaesthesiologists physical status I-III
* Elective Laparoscopic Cholecystectomy

Exclusion Criteria:

* Previous knowledge of difficult intubation
* Mouth opening less than 35 mm
* Cervical spine disease
* BMI≥35 kg/m2
* Upper respiratory or digestive tract disease
* Severe obstructive pulmonary disease
* Recent history of upper respiratory tract infection
* Pregnancy
* Patients who have a risk of gastric aspiration
* Preoperative sore throat
* Patients who refuse to participate

Withdrawal criterion:

-Orotracheal intubation during surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure pneumoperitoneum. | 10 month
  Oropharyngeal Leak Pressure (OLP) will be measured by closing the expiratory valve of the circle system at a fixed gas flow of 3 litres/min (maximum allowed 40 cmH2O) recording the pressure at which equilibrium has been reached or audible air is leaking.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa García-Navia, Principal Investigator — Hospital Plato
Locations (1):
- Anesthesia Department, Hospital Plató, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
All IPD that underlie results in a publication